CLINICAL TRIAL: NCT01883570
Title: Improving Search Strategy for Identifying Urgent Conditions on the Chest X-ray. (Original Title in French: Améliorer la stratégie de Recherche et l'Identification Des Conditions Urgentes Sur Une Radiographie Pulmonaire: Impact de l'Utilisation d'un Logiciel Interactif de Lecture systématique)
Brief Title: Improving Search Strategy for Identifying Urgent Conditions on the Chest X-ray
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CPER-11-120-D(1)
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Using Expert Visual Search Strategy to Train Students to Read the Chest X-ray
Keywords: visual search strategy, training, chest x-ray

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- trained visual search strategy (Experimental): An expert's visual search strategy for reading the chest x-ray was recorded using a gaze tracking device. This strategy was reproduced using a dynamic cursor and will be made available to participants in the experimental group using an interactive website.
  Interventions: Other: training in visual search strategy
- not trained in visual search strategy (Active Comparator): Participants will learn to read chest x-rays by having access to a library of chest x-rays identical to the one used by the experimental arm, but without the search strategy.
  Interventions: Other: access to a library of chest x-rays without search strategy

INTERVENTIONS:
Other: training in visual search strategy
  Arms: trained visual search strategy
Other: access to a library of chest x-rays without search strategy
  Arms: not trained in visual search strategy

SUMMARY:
Currently, teaching X-ray interpretation to medical students is not standardized, and is generally not very effective.

Objective: The goal of our study is to evaluate whether directly teaching an expert search strategy for x-ray interpretation to 3d year medical students is effective.

Methods:

* An expert's visual search strategy was recorded using a gaze-tracking device. The search strategy was then reproduced using a dynamic cursor moving across the corresponding chest x-ray, and incorporated into a teaching program accessible via the internet.
* Participants are 3rd year medical students who will be randomized into two groups. The experimental group will have access to the teaching program as described. The control group will have access to the same x-rays but not the expert's search strategy.
* At the end of the study period the investigators will collect performance data (the participants' accuracy at reading a series of chest x-rays) and process data (using gaze-tracking to evaluate the participants' search strategies); the experimental and control groups will be compared.

Expected results:

The investigators expect the group trained in expert search strategy to show improved accuracy at reading chest x-rays, and an improvement in their visual search strategy

ELIGIBILITY:
Inclusion Criteria:

* 3rd year medical students enrolled in medicine or surgery rotations during the planned study period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in medical student's visual search strategy at reading a chest x-ray | 2 months
  participants enrolled in the experimental group will be trained to learn the expert's search strategy for reading a chest x-ray. We hypothesize that by the end of the study period they will show an improved visual search strategy over students who were not trained in visual search but were taught through standard methods (interaction with clinician-educators during their clerkship rotations)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada